CLINICAL TRIAL: NCT05580757
Title: Role of Pharmacists in Suicide Prevention: Needs Assessment Among Pharmacists
Brief Title: Pharmacists as Gate Keepers in Suicide Prevention: Needs of Pharmacists
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0233
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Pharmacist-Patient Relations; Suicide; Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacists and pharmaceutical technical assistants (FTA): Dutch-speaking Belgian public pharmacists or pharmaceutical technical assistants (FTA)

SUMMARY:
This study aims to examine the opinions and needs of pharmacists and pharmaceutical technical assistants (FTA) concerning their role as gatekeepers in suicide prevention.

The primary objective is to map the experiences and needs of (public) pharmacists and FTA with regard to suicide prevention.

The secondary objective is to be able to develop more targeted tools, interventions or trainings based on the results of the needs assessment in order to facilitate the role of (public) pharmacists and FTA as gatekeepers in suicide prevention.

ELIGIBILITY:
Inclusion Criteria:

* Working as a (public) pharmacist or pharmaceutical technical assistant (FTA)
* 18 years or older
* Access to a computer, tablet or mobile phone with internet access
* Dutch-speaking

Exclusion Criteria:

* Hospital pharmacists or industrial pharmacists are not included in this study and thus constitute an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dutch-speaking Belgian public pharmacists or pharmaceutical technical assistants (FTA)
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Needs | Baseline. Completing the questionnaire will take approximately 15-20 minutes.
  Questionnaire based on a study by Gillette et al. (2020), scientific literature and previous needs surveys conducted by VLESP. In collaboration with the Flemish Pharmacists Network.
  Socio-demographics; Perceptions, attitudes and barriers: 55 statements (completely disagree, disagree, neutral, agree, completely agree); Contact with suicidal person (never/rarely, few times a year, monthly, weekly, daily), experience (very un-, rather un-, neutral, experienced, very experienced), possible actions as gatekeeper, referral, known organizations/helplines, previous education (yes or no), knowledge (yes/no)/ satisfaction (not at all, rather not, neutral, rather, very) existing education; Preparedness/need training (not at all, rather not, neutral, rather, very), preferred format of training, needed information; Suicidal thoughts/attempts (yes/no), hopelessness: 4 items (true/false)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No